CLINICAL TRIAL: NCT05942118
Title: A Monocentric, Prospective, Randomized Clinical Study Comparing ROLL (Radioguided Occult Lesion Localization) With Magnetic Markers for Preoperative Localization of Non-palpable Breast Lesions in Patients Undergoing Breast Conservative Surgery.
Brief Title: Comparison Between ROLL Versus Magnetic Seed for Preoperative Localization of Non-palpable Breast Lesion by Randomized Clinical Study.
Acronym: SEED02
Status: Recruiting | Type: Observational
Sponsor: Istituti Clinici Scientifici Maugeri SpA (Other)
Responsible Party: Principal Investigator, Fabio Corsi, Professor, Istituti Clinici Scientifici Maugeri SpA
Other Study IDs: 2778
Record Dates: First submitted 2023-06-23; First posted 2023-07-12 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer
Keywords: Non-palpable breast lesion
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- ROLL: Prior to surgery, an ultrasound-guided localization will be performed and albumin marked with Technetium 99m will be injected close to the tumor and in the subareolar area. During surgery, a specific probe will be used to locate the lesion and sentinel lymph node.
  Interventions: Procedure: Breast conservative surgery
- SEED: During diagnostic biopsy or prior to surgery, a magnetic clip will be placed in the breast lesion; during surgery, localization will be performed using a specific probe, while sentinel lymph node localisation, when needed, will be performed even with indocyanine green dye (ICG) or methylene blue dye
  Interventions: Procedure: Breast conservative surgery

INTERVENTIONS:
Procedure: Breast conservative surgery — Every patients with non-palpable breast lesion will undergo to conservative breast surgery after lesion's localization

SUMMARY:
Several localization techniques are now in use for localization of non-palpable breast lesions. Several studies have compared wire guided localization (WGL), which has been for years the gold standard for non-palpable breast lesions' localization, with more modern techniques. Scientific evidence supports the efficacy of the new "wire-free" techniques, which appear to be comparable to the WGL in terms of safe surgical resection, while overcoming limitations associated with logistic difficulties and patient discomfort. There is still limited data in literature on the comparative effectiveness of these modern techniques, and there is no strong evidence that one is superior to the others. In particular, no randomized trials of comparison between ROLL and magnetic seed localization are currently available. The aim of this randomized study is to compare ROLL with magnetic seed to assess their efficacy for non-palpable breast lesions' localization.

ELIGIBILITY:
Inclusion Criteria:

* Female;
* Non-palpable breast lesions;
* Indication to lesion's surgical excision (lumpectomy, quadrantectomy)
* Preoperative diagnosis on histology or cytology of borderline lesion (B3 or C3) or malignant lesion (B4-B5 or C4-C5);
* Written informed consent.

Exclusion Criteria:

* Benign lesion at diagnosis on preoperative core biopsy (B2) or fine needle aspiration (C2);
* Clinically palpable breast lesion;
* Breast lesion localization for planned neoadjuvant chemotherapy.

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Breast cancer patients with non-palpable lesions candidated for surgery
Sampling Method: Probability Sample
Enrollment: 262 (Estimated)
Dates: Start 2023-05-31 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Free-surgical margins | 3 years
  Number of surgical procedures in which surgical margins are disease-free ("no ink on tumor" for invasive cancer and margin of 2 mm for in situ-carcinoma).

SECONDARY OUTCOMES:
Excess breast resection | 3 years
  Excess breast resection calculated by the "calculated resection ratio" (CRR) as follow: CRR = total resection volume/optimal resection volume
Surgery Time | 3 years
  Surgery duration (hours)
Hospitalization days | 3 years
  Number of hospitalization's days
Complications | 3 years
  Complications occurred after biopsy or surgery
Reintervention | 3 years
  Reintervention rates
Cost-effectiveness analysis | 3 years
  Cost-effectiveness analysis in different subgroups
Follow up | 5 years after enrollment
  5-years follow-up outcomes

CONTACTS AND LOCATIONS:
Locations (1):
- Istituti Clinici Scientifici Maugeri SpA, Pavia, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No